CLINICAL TRIAL: NCT06713707
Title: Investigation of Validity and Reliability of the Minnesota Manual Dexterity Test in Patients with Parkinson's Disease
Brief Title: Investigation of Validity and Reliability of the Minnesota Manual Dexterity Test in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sefa Eldemir, Research Assistant, Cumhuriyet University
Other Study IDs: 7-PD-Minnesota-validity
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Minnesota manual dexterity; Validity; Reliability; upper limb function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Test Group: Patients with Parkinson's disease
  Interventions: Other: Manuel dexterity; Other: Manual Dexterity (only MMDT)
- Control Group: Healthy group
  Interventions: Other: Manual Dexterity (only MMDT)

INTERVENTIONS:
Other: Manuel dexterity — Individuals who meet the inclusion criteria will be evaluated for manual dexterity using 9-HPT, and JTHFT.
  Groups: Test Group
Other: Manual Dexterity (only MMDT) — Individuals who meet the inclusion criteria will be evaluated for manual dexterity using MMDT on a predetermined day.

SUMMARY:
Parkinson's Disease (PD) is a disease that affects upper extremity functional skills with clinical findings such as bradykinesia, rigidity, and hypokinesia, and causes limitations in patients' daily life activities. The impairment of upper extremity functional skills is related to the deficiency in planning both voluntary and complex movements, as well as the deficiency in multiple motor planning. In particular; fine manual dexterity, reaching, and grasping movements are affected, greatly affecting patients' daily activities. Therefore, upper extremity evaluations are an important issue to consider for training upper extremity motor skills in PD. There are minimal assessment tools for evaluating the upper extremity functions of individuals with PD. The Nine-Hole Peg Test and the Jebsen Hand Function Evaluation Test are the most commonly used scales in the evaluation of the upper extremity in PD, and their validity and reliability have been demonstrated. These scales roughly evaluate both extremities separately. However, these scales are not suitable assessment tools for testing activities in which both extremities are frequently used in daily life. Therefore, there is a need for valid and reliable scales that can evaluate upper extremity activities both in isolation and bilaterally. The Minnesota manual dexterity test (MMDT) allows both hands to be evaluated together. It also evaluates hand-eye coordination and gross motor skills in addition to manual dexterity. MMDT is used in individuals with PD, but there is no study in the literature examining the validity and reliability of the scale. Therefore, this study aims to evaluate the reliability and validity of MMDT in individuals with PD.

DETAILED DESCRIPTION:
At baseline, the MMDT, 9-hole peg test, and Jebsen-Taylor Hand Function Test (JTHFT) will be applied to the MS group. The MMDT will be repeated seven days after the first application in MS. Healthy controls are going to perform only the MMDT.

ELIGIBILITY:
Inclusion Criteria:

* Between 40-80 years old
* Diagnosed with only "Parkinson's Disease" by a neurologist
* Between 1-3 values of your thoughts according to Hoehn and Yahr manufacturers

Exclusion Criteria:

* Having any vision, hearing or perception problems that may affect the research results,
* Having an orthopedic problem that may affect manual skills in the upper extremity,
* Having a cardiovascular, pulmonary disorder

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease who apply to Sivas Cumhuriyet University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Minnesota Manual Dexterity Test | baseline (on the predetermined assessment day)
  The Minnesota Manual Dexterity Test (MMDT) is a performance test designed to evaluate hand functions and hand-eye coordination both unilaterally and bilaterally, higher scores mean a worse outcome
Minnesota Manual Dexterity Test-second | the second assessment will be conducted after the one week
  The Minnesota Manual Dexterity Test (MMDT) is a performance test designed to evaluate hand functions and hand-eye coordination both unilaterally and bilaterally, higher scores mean a worse outcome

SECONDARY OUTCOMES:
9-Hole Peg Test | baseline (on the predetermined assessment day)
  The 9-Hole Peg Test (9-HPT) evaluates hand dexterity based on performance, higher scores mean a worse outcome
The Jebsen Hand Function Test | baseline (on the predetermined assessment day)
  The Jebsen Hand Function Test (JHFT) is one of the objective and standardized tests that assesses fine motor skills and functional hand use by simulating daily living activities, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas/Center, Turkey (Türkiye)

REFERENCES:
- [Background] Earhart GM, Cavanaugh JT, Ellis T, Ford MP, Foreman KB, Dibble L. The 9-hole PEG test of upper extremity function: average values, test-retest reliability, and factors contributing to performance in people with Parkinson disease. J Neurol Phys Ther. 2011 Dec;35(4):157-63. doi: 10.1097/NPT.0b013e318235da08. PMID 22020457
- [Background] Mak MK, Lau ET, Tam VW, Woo CW, Yuen SK. Use of Jebsen Taylor Hand Function Test in evaluating the hand dexterity in people with Parkinson's disease. J Hand Ther. 2015 Oct-Dec;28(4):389-94; quiz 395. doi: 10.1016/j.jht.2015.05.002. Epub 2015 May 18. PMID 26227308
- [Background] Ovacik U, Tarakci E, Gungor F, Menengic KN, Leblebici G, Acar ZO, Soysal A. The minnesota manual dexterity test as a bimanual performance measure in people with multiple sclerosis. Mult Scler Relat Disord. 2022 Aug;64:103943. doi: 10.1016/j.msard.2022.103943. Epub 2022 Jun 6. PMID 35738113